CLINICAL TRIAL: NCT07221448
Title: Improving Vascular Health Using Nutrition Education Aimed At Increasing Potassium Intake Versus Reducing Sodium Intake
Brief Title: Sodium vs Potassium Education to Improve Vascular Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrea Lobene, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005997; 2025-67017-44996 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: sodium; potassium; nutrition education; endothelial function; cardiovascular disease risk factors
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High potassium dietary education (Experimental)
  Interventions: Behavioral: High potassium dietary education/counseling
- Low sodium dietary education (Active Comparator)
  Interventions: Behavioral: Low sodium dietary education/counseling

INTERVENTIONS:
Behavioral: High potassium dietary education/counseling — Participants assigned to this intervention arm will receive four weekly individualized education sessions on how to increase their dietary potassium intake.
  Arms: High potassium dietary education
Behavioral: Low sodium dietary education/counseling — Participants assigned to this intervention arm will receive four weekly individualized education sessions on how to reduce their dietary sodium intake.
  Arms: Low sodium dietary education

SUMMARY:
The goal of this clinical trial is to determine if a self-selected high potassium diet is easier to achieve and more effective at improving vascular health than a low sodium diet in generally healthy young adults who typically consume more than the recommended amount of sodium. The main questions it aims to answer are:

1. Is it easier for young adults to increase their potassium intake, rather than reduce their sodium intake?
2. Is a self-selected high potassium diet better at improving vascular health compared to a self-selected low sodium diet?

Researchers will compare the effectiveness of an education-based intervention centered only on increasing dietary potassium intake against an education-based intervention centered only on reducing dietary sodium intake.

Participants will be randomly assigned to receive comprehensive dietary education on adopting either a high-potassium diet or a low-sodium diet.

Education will be delivered in four weekly one-on-one sessions. Following the four-week education period, participants will be encouraged to change their diet based on what they have learned. Measures of dietary compliance (urine samples and diet records) and cardiovascular health (blood pressure, endothelial function) will be assessed at two, four, and six months post-education.

DETAILED DESCRIPTION:
High sodium diets are a major contributor to cardiovascular disease. Unfortunately, reducing sodium intake can be challenging. It is known that increasing potassium intake can improve cardiovascular disease risk factors in a laboratory setting. The investigators are hoping to show that it is more feasible and effective for individuals to increase their potassium intake, rather than reduce their sodium intake, to improve cardiovascular disease risk factors, including blood pressure and endothelial function.

In this study, participants will be randomly assigned to receive individualized education over the course of four weeks to help them adopt one of two dietary patterns: 1) a self-selected low sodium diet (goal: ≤1,500 mg/day) or 2) a self-selected high potassium diet (goal: ≥4,700 mg/day). Participants will be provided individualized nutrition education once per week, at the participant's convenience by trained study staff to help them meet the target nutrition goals. No food, supplements, or devices will be provided to participants, and participants will be advised not to take any dietary supplements containing potassium during the intervention and follow-up period. Follow up with participants will be every two months for six months post-education to measure compliance with the desired dietary changes as well as changes in cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend in-person laboratory visits
* Usual sodium intake ≥3,000 mg/d for females and ≥4,000 mg/d for males
* Usual potassium intake ≤2,500 mg/d in females and ≤3,000 mg/d in males

Exclusion Criteria:

* BMI ≥35 kg/m2
* Seated blood pressure ≥130/80 mmHg
* Current diagnosis or history of diabetes, renal disease, cancer, cardiovascular disease, or major cardiovascular event (e.g. heart attack or stroke)
* Current or recent use of a diuretic (within the past 6 months)
* Elevated blood lipids (LDL cholesterol ≥190 mg/dL)
* Elevated serum potassium level (>5.1 mmol/L)
* Elevated BUN (>22 mg/dL)
* Elevated creatinine (>1.2 mg/dL)
* Low eGFR (<90 mL/min/1.73 m²)
* Current or recent use of tobacco, nicotine, or illicit drugs
* Radical hysterectomy or oophorectomy (females)*
* Pregnant or lactating
* Following a weight-loss diet, or intending to gain or lose weight during the study period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in dietary sodium intake | Baseline; 2 month, 4month, 6month
  Dietary sodium intake will be assessed via participant self-reported 3 day diet record
Change in dietary potassium intake | Baseline, 2month, 4month, 6month
  Dietary potassium intake will be assessed via participant self-reported 3-day diet record
Change in 24-hour urinary sodium excretion | Baseline, 2month, 4month, 6month
  Urinary sodium excretion obtained from 24-hour urine sample
Change in 24-hour urinary potassium excretion | Baseline, 2month, 4month, 6month
  Urinary potassium excretion measured from 24-hour urine sample
Change in Blood pressure | Baseline; 2 month, 4month, 6month
  Seated, automated blood pressure mmHg
Change in Endothelial function | Baseline; 2 month, 4month, 6month
  brachial artery flow-mediated dilation as measured in % dilation

SECONDARY OUTCOMES:
Direct measurement of arterial stiffness | Baseline, 2month, 4month, 6month
  Carotid-femoral pulse wave velocity reported in m/s
Indirect measurement of arterial stiffness | Baseline, 2month, 4month, 6month
  Augmentation obtained from the brachial artery pressure waveform using a blood pressure cuff on the upper arm, reported as %

OTHER OUTCOMES:
Change in Body weight | Baseline; 2 month, 4month, 6month
  body weight assessed in kilograms
Change in total cholesterol | Baseline, 2month, 4month, 6month
  Fasting total cholesterol obtained as part of standard lipid panel
Change in LDL cholesterol | Baseline, 2month, 4month, 6month
  Fasting LDL cholesterol obtained as part of a standard lipid panel
Change in HDL cholesterol | Baseline, 2month, 4month, 6month
  Fasting HDL cholesterol obtained as part of a standard lipid panel
Change in triglycerides | Baseline, 2month, 4month, 6month
  Fasting triglycerides obtained as part of a standard lipid panel

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lobene, PhD, RD, LD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No